CLINICAL TRIAL: NCT07151092
Title: Exploring Experiences of Adolescent Suicide Loss Survivors After Participating in a Grief Intervention Group
Brief Title: Adolescent Suicide Loss Survivors Grief Intervention Group
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Carly Paro, Associate Professor, Nova Southeastern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-390
Record Dates: First submitted 2025-08-27; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Grief
Keywords: Suicide Loss; Stigmatized Grief; Bereavement; Traumatic grief; adolescent grief group; coping; continuing bonds; hope
MeSH Terms: conditions — Prolonged Grief Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adolescent Grief Group (Experimental): Participants will include up to 20 adolescents (ages 13-17) who are survivors of suicide loss and have volunteered to participate in the one day experiential group intervention that will include education, interaction, and client centered counseling groups.
  Interventions: Behavioral: Adolescent Grief Group

INTERVENTIONS:
Behavioral: Adolescent Grief Group — The intervention will include psycho-education, peer-support, and professional supportive counseling from licensed clinicians.

SUMMARY:
This study will provide evidence-based recommendations for designing interventions tailored to adolescents dealing with suicide loss. By exploring how these young people experience and make meaning of their grief, the study will contribute to the development of best practices for mental health professionals and educators working with suicide loss survivors. This study will provide evidence-based recommendations for designing interventions tailored to adolescents dealing with suicide loss. By exploring how these young people experience and make meaning of their grief, the study will contribute to the development of best practices for mental health professionals and educators working with suicide loss survivors.

This study will enhance scientific understanding by examining how adolescents experience grief after suicide loss and identifying which components of bereavement interventions are most effective for this age group. It will improve societal welfare by informing the development of targeted, evidence-based support programs that address the unique mental health needs of bereaved adolescents. Long-term, the findings may reduce the risk of complicated grief and suicidality, support emotional resilience, and guide best practices in schools, clinics, and community settings for supporting youth after traumatic loss.

DETAILED DESCRIPTION:
This study will provide evidence-based recommendations for designing interventions tailored to adolescents dealing with suicide loss. By exploring how these young people experience and make meaning of their grief, the study will contribute to the development of best practices for mental health professionals and educators working with suicide loss survivors. This study will provide evidence-based recommendations for designing interventions tailored to adolescents dealing with suicide loss. By exploring how these young people experience and make meaning of their grief, the study will contribute to the development of best practices for mental health professionals and educators working with suicide loss survivors. It is hypostasized that the results from this study will show significant impact in the areas of hope, healthy coping, grief, continuing bonds, and connection. In additional it will create support systems for these teens that promote mental health and reduce the risk of long-term psychological consequences associated with suicide loss.

The procedure for this study is as follows:

1. Recruitment and Consent (One Time)

   Procedure: Community partners will assist with recruitment through social media, community events, and collaboration with local mental health agencies.

   Initial Contact: Any potential participants and their guardians who contact the PI or Co-PI will attend an information session conducted via Zoom or phone call prior to being consent.

   Consent Process: Prior to starting the group session potential participants and their guardians will be consented. Researchers will explain the study and review consent and assent forms. Time will be allotted for questions.
2. Pretest Survey (One Time)

   Instruments Administered:

   Demographic Survey (custom) will be included before starting the other measures Hogan Inventory of Bereavement - Short Form, Child and Adolescent (HIB-SF-CA) Brief COPE Inventory (BCI) Continuing Bonds Scale (CBS) Perceived Hope Scale (PHS)
3. Day-of Intervention (One Time Event)

   Prior to starting the group intervention the participants will be given a brief intake to better understand their personal relationship to their loss.

   Structure: 4-hour single-day grief group intervention broken down into the following parts:

   Part 1 : Intake Survey, Guest speaker presentation on grief and coping with journal reflection Part 2 : Viewing of AFSP video on suicide loss + guided discussion Part 3 : Therapeutic process group facilitated by licensed clinicians Part 4 : Artistic expression and closing activity
4. After the Intervention participants will be given a posttest and participate in a focus group.

   Assessment to be given after the intervention include the Therapeutic Factors Inventory - Short Form (TFI-S) administered via iPads Focus group interview about the participant's experience of the workshop
5. Two-Week after the Intervention there will be a follow-up focus group, and the following instruments will be administered:

   Instruments Administered:

   HIB-SF-CA Brief COPE Inventory Continuing Bonds Scale Perceived Hope Scale
6. Six-Weeks after the intervention there will be a follow-up focus group and the following instruments will be administered:

Instruments Administered:

HIB-SF-CA Brief COPE Inventory Continuing Bonds Scale Perceived Hope Scale

The research that guided this study are stated below.

Overarching Mixed Methods Question:

How do the experiences of adolescent suicide loss survivors help explain the adolescent's grief, personal growth, hope, coping, and ongoing connections with deceased loved ones after an interactive grief group intervention?

Overarching Quantitative Research Question:

How does an interactive grief group intervention affect adolescent suicide loss survivors' experiences of grief, personal growth, hope, coping, and ongoing connections with deceased loved ones?

Quantitative subquestions:

1. How does participation in an interactive grief group intervention affect adolescent suicide survivors' grief experiences, as measured by the Hogan Inventory of Bereavement?
2. How does participation in an interactive grief group intervention influence participants' personal growth, as assessed by the Hogan Inventory of Bereavement?
3. How does the level of hope, as measured by the Perceived Hope Scale, change for participants after engaging in the interactive grief group intervention?
4. How does participation in the interactive grief group intervention impact adaptive coping strategies, as measured by the Brief COPE inventory?
5. How does the interactive grief group intervention affect ongoing connections with the deceased, as measured by the Continuing Bonds Scale?
6. How do therapeutic group factors, as measured by the Therapeutic Factors Inventory for Groups (TFI-S), correlate with hope, coping, grief, and personal growth post-intervention?

Hypothesis

Hypothesis 1a: Participation in an interactive grief group intervention will significantly reduce grief experiences among adolescent suicide loss survivors, as measured by the Hogan Inventory of Bereavement.

Hypothesis 1b: Participation in an interactive grief group intervention will significantly increase personal growth among adolescent suicide loss survivors, as measured by the Hogan Inventory of Bereavement.

Hypothesis 1c: Participation in an interactive grief group intervention will significantly increase participants' hope, as measured by the Perceived Hope Scale.

Hypothesis 1d: Participation in an interactive grief group intervention will significantly increase participants' adaptive coping strategies, as measured by the Brief COPE inventory.

Hypothesis 1e: Participation in an interactive grief group intervention will significantly increase ongoing connections with the deceased, as measured by the Continuing Bonds Scale.

Hypothesis 1f: There will be a significant positive correlation between the therapeutic factors (as measured by the Therapeutic Factors Inventory for Groups - TFI-S) and participants' hope, coping, grief, and personal growth post-intervention.

Overarching Qualitative Research Question: These questions will be guided using an interview protocol for the focus groups.

How do suicide loss survivors experience an interactive grief group intervention?

Qualitative Subquestions:

1. How do participants articulate and understand their grief experiences after the group intervention?
2. In what ways do participants express their experiences of personal growth following the group intervention?
3. How do participants perceive and articulate the role of hope in their lives following the group intervention?
4. How do participants describe their coping mechanisms and adaptations after experiencing the group intervention?
5. How do participants perceive their ongoing connections with the deceased after the group intervention?
6. How do participants describe the group experience as a whole?
7. How do they experience their facilitators, the other members of the group?

ELIGIBILITY:
Inclusion Criteria:

* - Adolescents aged 13-17 years.
* Survivor of suicide loss.
* Permission from parent or guardian.

Exclusion Criteria:

* Adolescents who have not experienced the loss of a loved one to suicide.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Hope & Coping | Pre intervention, 2 weeks post, 6 weeks post
  Perceived Hope Scale and Brief COPE
Grief Experience | Pre intervention, 2 weeks post, and 6 weeks post.
  Hogan Inventory of Bereavement, Short Form, Child and Adolescent HIB-SF-CA
Continuing Bonds | Pre-intervention, 2 weeks post, 6 weeks post intervention
  Continuing Bonds Scale
Personal Growth | Pre intervention, 2 weeks post, 6 weeks post
  the Hogan Inventory of Bereavement, Short Form, Child and Adolescent HIB-SF-CA
Therapeutic Factors | Immediately following Intervention
  Therapeutic Factors Inventory- Short Form TFI-S

IPD SHARING:
Plan to Share IPD: No